CLINICAL TRIAL: NCT03820193
Title: Traditional vs. Nonopioid Analgesia After Arthroscopic Meniscus Surgery
Brief Title: Nonopioid Analgesia After Arthroscopic Meniscus Surgery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Charles S Day, Orthopedic Surgeon, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 123193
Record Dates: First submitted 2019-01-25; First posted 2019-01-29 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Meniscus Disorder; Narcotic Use
MeSH Terms: interventions — Celecoxib; Hydrocodone; Acetaminophen; oxycodone-acetaminophen; Ketorolac; Ketorolac Tromethamine; Gabapentin; Diazepam

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Post-Operative Non Opioid Pain Protocol (Experimental): Patients will be administered a post-operative non-opioid pain protocol consisting of: Celecoxib, Ketorolac, Gabapentin, Acetaminophen, Diazepam
  Interventions: Drug: Celecoxib; Drug: Ketorolac; Drug: Gabapentin; Drug: Acetaminophen; Drug: Diazepam
- Post-Operative Traditional Pain Protocol (Active Comparator): Patients will be administered a traditional post-operative pain protocol consisting of: Hydrocodone-acetaminophen
  Interventions: Drug: Hydrocodon/Acetaminophen

INTERVENTIONS:
Drug: Celecoxib — Post-Operative Non Opioid Pain Protocol
  Other Names: Celebrex
  Arms: Post-Operative Non Opioid Pain Protocol
Drug: Hydrocodon/Acetaminophen — Traditionally used narcotic pain control
  Other Names: Norco
  Arms: Post-Operative Traditional Pain Protocol
Drug: Ketorolac — Post-Operative Non Opioid Pain Protocol
  Other Names: Toradol
  Arms: Post-Operative Non Opioid Pain Protocol
Drug: Gabapentin — Post-Operative Non Opioid Pain Protocol
  Other Names: Neurontin
  Arms: Post-Operative Non Opioid Pain Protocol
Drug: Acetaminophen — Post-Operative Non Opioid Pain Protocol
  Other Names: Tylenol
  Arms: Post-Operative Non Opioid Pain Protocol
Drug: Diazepam — Post-Operative Non Opioid Pain Protocol
  Other Names: Valium
  Arms: Post-Operative Non Opioid Pain Protocol

SUMMARY:
This is a randomized, single blinded, standard of care controlled clinical trial. This project aims to compare postoperative pain control in patients in two treatment arms of arthroscopic meniscus surgery: a treatment group given a non-opioid pain control regimen, and a standard of care control group given standard opioid pain control regimen

DETAILED DESCRIPTION:
Study Design: This is a randomized, single blinded, standard of care-controlled clinical trial. All adult patients over eighteen desiring arthroscopic meniscus surgery will be eligible. Nonnarcotic postoperative pain control regimen described below were chosen based on previous studies in fracture care and joint arthroplasty.

Patients will be consented and recruited. Once participation has been determined and consent obtained, the names of participating patients will be provided to the research pharmacy. Patients will be randomized with a computer-generated table in 2 patient blocks by the research pharmacy. Patients postoperative analgesia will be divided into one of the following 2 treatment arms: 1) A novel nonopioid pain protocol or 2) traditional narcotic pain analgesia

Primary endpoints is reduction in pain as measured by Visual Analog Score and Patient Reported Outcome Measurement Informatics Systems. The endpoints will be collected at each post-operative day using a journal. Moreover, endpoints will be collected at the patient's first post-operative appointment. These appointments are scheduled within one-week of the index procedure.

Statistical Analysis: All continuous data will be analyzed using independent 2-group t tests and reported as means ± standard deviations. Categorical data will be compared between the 2 groups using chi-square tests and reported as counts and percentages. A preliminary test to confirm the quality of variances will be conducted prior to utilizing the t test to confirm the appropriate statistical analysis. Nonparametric equivalents Wilcoxon rank-sum and Fisher exact tests will be used as needed for nonnormal distributions and low variable numbers, respectively. A multivariable regression analysis was performed to assess for potential confounding demographic variables.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients over age 18 scheduled for arthroscopic meniscus repair or partial menisectomy

Exclusion Criteria:

* Patients with a medical history of known allergies or intolerance to allergies or intolerance to Celebrex, Tylenol, Neurontin, dexamethasone, tramadol, substantial alcohol or drug abuse, and pregnancy, history of narcotics within 6 months of surgery, renal impairment, peptic ulcer disease, GI bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Pain Levels | 10 days post-operatively
  Patients record pain levels every 3 hours using Visual analog scales for 10 days post-operatively. Average daily pain was calculated for each patient. Higher values portend worse control.
Patient Reported Outcome Measurement Information System | 10 days post-operatively
  Patient Reported Outcome Measurement Information System - Pain Interference (PROMIS PI) scores collected nightly until study completion. Average PROMIS PI values calculated nightly. A higher score indicates more pain interference.

CONTACTS AND LOCATIONS:
Overall Officials: Toufic R Jildeh, MD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided
Per Request